CLINICAL TRIAL: NCT03498209
Title: Prevalence of Molar Incisor Hypominerlization (MIH) Among a Group of Egyptian Children: A Cross Sectional Study
Brief Title: Prevalence of Molar Incisor Hypominerlization (MIH) Among a Group of Egyptian Children
Acronym: MIH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, shahinda abdeen, Dr.shahinda abdeen pedodontist principal investigator, Cairo University
Other Study IDs: prevalence of MIH
Record Dates: First submitted 2018-04-07; First posted 2018-04-13 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the Prevalence of MIH in a group of Egyptian children attending the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University.

DETAILED DESCRIPTION:
One single operator, Master degree student in the department of Pediatric Dentistry and Dental public health, Faculty of Dentistry, Cairo University will assess incidence of molar incisor hypomineralization for all the patients who will be included in the study sample. The survey will involve a structured questionnaire which will be followed by clinical examination to assess the presence / absence of molar incisor hypomineralization and its severity based on EAPD criteria

ELIGIBILITY:
Inclusion Criteria:

1. Children age from eight to twelve years.
2. Medically free.
3. Singed informed consent.
4. Both sexes are included
5. Parent and children cooperation.

Exclusion Criteria:

1. Children with (amelogenesis imperfecta, tetracycline tooth stains, extensive destruction due to caries, or have restoration or crown and fluorosis).
2. Children with orthodontic bands on the first permanent molars preventing adequate clinical examination.

Ages: 8 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Data for this study will be conducted in Department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University, Egypt.
  Participants will be selected from the outpatient's clinic of Pediatric Dentistry and Dental Public Health department, Faculty of Dentistry, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-20 (Estimated); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of molar incisor hypomineralization among a group of Egyptian Children | baseline
  prevalence of molar incisor hypomineralization measured by clinical examination

SECONDARY OUTCOMES:
Relationship of MIH with dental caries | baseline
  Relationship of MIH with dental caries measured by caries index

CONTACTS AND LOCATIONS:
Overall Officials: eman S ELMASRY, PHD, Study Director — Cairo University

REFERENCES:
- [Background] Biondi AM, Lopez Jordi Mdel C, Cortese SG, Alvarez L, Salveraglio I, Ortolani AM. Prevalence of molar-incisor hypomineralization (MIH) in children seeking dental care at the Schools of Dentistry of the University of Buenos Aires (Argentina) and University of la Republica (Uruguay). Acta Odontol Latinoam. 2012;25(2):224-30. PMID 23230646
- See also: Prevalence of molar incisor hypomineralization in school children aged 8-12 years in Chennai — http://www.jisppd.com/article.asp?issn=0970-4388;year=2016;volume=34;issue=2;spage=134;epage=138;aulast=Yannam